CLINICAL TRIAL: NCT04274608
Title: Intra-gastric Fundal and Body Injection of Botulinum Toxin A for Weight Loss, a Randomized Controlled Trial
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Danson Yeo Xue Wei, Associate Consultant, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TanTockSengH
Record Dates: First submitted 2020-02-16; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Patients in the intervention arm will receive 300units of Botulinum Toxin A (Botox; Allergan Inc., Irvine, Ca, USA) diluted to 10mls of saline. Endoscopy will be performed using a single-lumen gastroscope. Injection of the solution will be done using a 23Gauge Interject needle catheter. 20 separate injections of 0.5ml each will be performed in a concentric ring 1cm apart. 10 injections will be performed into the body of the stomach, and 10 injections into the fundus, from the level of the CEJ and above
  Patients will undergo a 12-week weight management program approximately 2 weeks after the injection of Botox.
  Interventions: Drug: Botulinum toxin type A; Behavioral: Weight Management Program
- Control Arm (Active Comparator): Patients will undergo a 12-week weight management program.
  Interventions: Behavioral: Weight Management Program

INTERVENTIONS:
Drug: Botulinum toxin type A — Intragastric injection of Botulinum toxin type A
  Arms: Intervention Arm
Behavioral: Weight Management Program — 12 week weight management program

SUMMARY:
This is a randomized controlled trial to compare intra-gastric injection of Botulinum Toxin A (Botox; Allergan Inc. Irvine, Ca, USA) against non-surgical management for obesity (i.e. exercise/diet). Our hypothesis is that intra-gastric injection of Botox into the fundus and body of the stomach will result in greater weight loss than just exercise and diet alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 to 65yrs old
2. BMI >32.5 (Class II obesity)

Exclusion Criteria:

1. Pregnancy or lactation
2. Known pre-existing neuromuscular disorders or peripheral motor neuropathic disease (e.g. amyotrophic lateral sclerosis, motor neuropathy)
3. Patients with known liver cirrhosis or known esophageal/gastric varices
4. Known eating disorders
5. Known major cardiovascular or pulmonary conditions
6. Previous gastric/bariatric surgery
7. Pathologic changes of the esophagus/stomach/duodenum demonstrated on endoscopy (esophagitis, peptic ulcers, cancer)
8. Known alcohol or drug abuse
9. Known allergy to any ingredients in Botox or allergic reaction to any other botulinum toxin product

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 1 year
  Examine the average weight loss
Time to weight regain following a single injection of intra-gastric Botox | 1 year

SECONDARY OUTCOMES:
Gut hormone level | 1 year
  Ghrelin
Gut hormone level ( Leptin) | 1 year
  Leptin
Satiety index | 1 year
Co-morbidities | 1 year
  Diabetes, hypertension, hyperlipidemia

CONTACTS AND LOCATIONS:
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore